CLINICAL TRIAL: NCT04903197
Title: A Phase Ib, Multi-center, Open-label Dose Escalation and Expansion Platform Study of VAY736 as Single Agent and in Combination With Select Antineoplastic Agents in Patients With Non-Hodgkin Lymphoma (NHL)
Brief Title: Study of VAY736 as Single Agent and in Combination With Select Antineoplastic Agents in Patients With Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision and not due to any safety or tolerability concerns.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CVAY736J12101; 2020-005881-32 (EudraCT Number)
Record Dates: First submitted 2021-05-25; First posted 2021-05-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Non-Hodgkin Lymphoma, Diffuse Large B Cell Lymphoma, Follicular Lymphoma, Mantle Cell Lymphoma, Marginal Zone Lymphoma
Keywords: VAY736; ianalumab; lenalidomide; non-Hodgkin lymphoma; NHL; Diffuse large B cell lymphoma; DLBCL; Follicular lymphoma; FL; Mantle cell lymphoma; MCL; Marginal zone lymphoma; MZL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — ianalumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1A (Experimental): VAY736 single agent dose escalation in patients with NHL subtypes of diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL)
  Interventions: Drug: VAY736
- Arm 1B (Experimental): VAY736 single agent dose expansion in patients with DLBCL. This arm was not conducted.
  Interventions: Drug: VAY736
- Arm 2A (Experimental): VAY736 + lenalidomide dose escalation in patients with DLBCL, follicular lymphoma (FL), mantle cell lymphoma (MCL) and marginal zone lymphoma (MZL).
  Interventions: Drug: VAY736; Drug: lenalidomide
- Arm 2B (Experimental): VAY736 + lenalidomide dose expansion in patients with DLBCL. This arm was not conducted.
  Interventions: Drug: VAY736; Drug: lenalidomide

INTERVENTIONS:
Drug: VAY736 — VAY736 is a fully human IgG1 monoclonal antibody (mAb) which targets the B cell activating factor receptor (BAFF-R) expressed on the surface of differentiated B cells and modulates their function.
  Other Names: ianalumab
Drug: lenalidomide — Immune-modulatory agent that enhances activation of NK cells.
  Arms: Arm 2A; Arm 2B

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics (PK), immunogenicity and preliminary efficacy of VAY736 alone or in combination with other therapies in patients with NHL in a platform trial.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the safety and tolerability in patients with NHL and identify a maximum tolerated dose (MTD) and/or recommended dose (RD) of VAY736 single agent and in combination with other anti-cancer therapies.

This is a phase I/Ib, multi-center, open-label study with multiple treatment arms in an adaptive study design. The study is comprised of a dose escalation part and dose expansion part.

In dose escalation, the investigational drug VAY736 was explored alone or in combination with lenalidomide. Increasing doses of VAY736 alone or in combination were given to small groups of patients to identify the maximum tolerated dose/recommended dose (MTD/RD) in patients with NHL. In dose expansion, some or all the treatments from dose escalation could be tested at the recommended doses in patients with NHL. The study was expected to last approximately 4 years (from the enrollment of the first patient to the discontinuation of the last patient), but it was terminated early due to a business decision, not because of any safety or tolerability concerns. Consequently, the dose expansion part was not conducted.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with confirmed diagnosis of relapsed/refractory B-cell NHL with all subtypes of DLBCL, follicular lymphoma (FL), marginal zone lymphoma (MZL) and mantle cell lymphoma (MCL) per WHO 2016 criteria. Patients in subtype arm e.g. DLBCL must have confirmed diagnosis of relapsed/refractory DLBCL.
* Received and failed or be intolerant to standard of care therapy (at least two prior lines, including an anti-CD20 therapy for NHL)
* Must have measurable disease and ECOG of 0 to 2

Exclusion Criteria:

* Baseline laboratory results outside of protocol defined ranges
* Patients with primary CNS lymphoma
* History of hypersensitivity to VAY736 or any drugs in similar chemical classes (e.g. monoclonal antibodies)
* Impaired cardiac function or clinically significant cardiac disease
* History of or current interstitial lung disease or pneumonitis grade 2 or higher
* HIV infection
* Active hepatitis C infection and/or hepatitis B infection
* Pregnant or nursing (lactating) women
* Women of child-bearing potential unless they are using highly effective methods of contraception

Other Inclusion/Exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of dose limiting toxicities (DLTs) | 28 days (first cycle of treatment)
  Safety and tolerability
Incidence of Adverse events (AEs) and serious adverse events (SAEs) | 4 years
  Incidence of AEs and SAEs is defined as number of participants with AEs and SAEs, including changes from baseline in vital signs, electrocardiograms (ECGs) and laboratory results qualifying and reported as AEs.
Number of patients with dose interruptions and dose reductions | 4 years
  Safety and tolerability
Dose intensity | 4 years
  Safety and tolerability

SECONDARY OUTCOMES:
Overall response rate (ORR) | 4 years
  Efficacy will be assessed by Lugano Classification (FDG-PET/CT scans)
Best overall response (BOR) rate | 4 years
  Efficacy will be assessed by Lugano Classification (FDG-PET/CT scans)
Area under curve (AUC) for VAY736 and combination partners | 4 years
  PK parameters will be derived from serum concentrations
Maximum observed drug concentration after single dose administration (Cmax) for VAY736 and combination partners | 4 years
  PK parameters will be derived from serum concentrations
Change from baseline in anti-drug antibodies (ADA) | Baseline, 4 years
  Blood samples will be collected to detect change in levels of antibodies to VAY736

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Institutes of Biomedical Research, Study Director — Novartis Institutes of Biomedical Research
Locations (9):
- Novartis Investigative Site, Melbourne, Victoria, Australia
- China (2):
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Novartis Investigative Site, Leipzig, Germany
- Italy (2):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Rozzano, MI
- Novartis Investigative Site, Yamagata, Japan
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CVAY736J12101 Clinical Trial Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18405